CLINICAL TRIAL: NCT04693754
Title: Endoscopic Ultrasound Radiofrequency Ablation, Database Repository
Acronym: EUS-RFA
Status: Enrolling by invitation | Type: Observational
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, John DeWitt, Principal Invstigator, Indiana University
Other Study IDs: 2006385412
Record Dates: First submitted 2020-07-16; First posted 2021-01-05 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-01

CONDITIONS: Pancreatic Neoplasm
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The purpose of having this database is to collect data related to endoscopic ultrasound RFA procedures performed by Indiana University EUS physicians for the treatment of tumors or adenopathy. This database is a repository database only, all information will be obtained in the electronic medical record. No additional clinical procedures will be performed outside current standard of care for endoscopic ultrasound. The patient will have already signed an informed consent for the endoscopic ultrasound. Subjects will be entered into the database for up to 10 years after the most recent procedure.

DETAILED DESCRIPTION:
Radiofrequency ablation (RFA) is a well-established therapeutic option for ablation of dysplastic and neoplastic tissue by the use of local thermal coagulative necrosis. Options for administration include percutaneous or a surgical approach. Percutaneous RFA is effective and safe, but it is unfeasible in cases of lesions with interposition of organs and/or vessels. For lesions such as the pancreas, surgery-assisted RFA has been described but requires general anesthesia and is associated with a substantial risk of thermal injuries to major vessels or adjacent structures.

EUS-guided RFA is a minimally invasive approach that offers high-quality real-time imaging guidance during selective ablation of benign (1-5) or malignant (6-7) pancreatic lesions. Treatment in small case series has shown to produce local necrosis with minimal adverse events. Other sites treated include the liver and metastatic adenopathy.

This database will collect data related to endoscopic ultrasound RFA procedures performed by Indiana University EUS physicians for the treatment of tumors or adenopathy. No additional clinical procedures will be performed outside current standard of care for endoscopic ultrasound. The patient's information collected will be pre-procedure identification of the adenopathy, labs, the endoscopic ultrasound(s) and post procedure follow up and care related to the adenopathy.

Patients will be contacted by phone at post-procedure 1 & 2 weeks and asked to report symptoms related to the procedure.

ELIGIBILITY:
Inclusion Criteria:

Subjects 14 years of age and older Referral for the treatment of a benign or malignant tumor or adenopathy

Exclusion Criteria:

* Subjects less than 14 years of age Unable to comprehend the study consent due to language or disability

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Above 14 years of age and referred for treatment of benign or malignant tumor or adenopathy
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of any procedural complications that occur during the procedure on date of procedure. | Day of procedure
  This data will be used for to determine the clinical impact and safety of these procedures.
Rate of patient report of symptoms related to procedure (Acute pancreatitis, abdominal pain, infection/abscess, venous thrombosis, & fever) | 1 week following procedure
  1 week phone follow up
Rate of patient report of symptoms related to procedure (Acute pancreatitis, abdominal pain, infection/abscess, venous thrombosis, & fever) | 2 weeks following procedure
  2 week phone follow up

CONTACTS AND LOCATIONS:
Locations (1):
- Indiana University Health University Hospital, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No